CLINICAL TRIAL: NCT02337517
Title: Pilot Study for the Treatment of Steroid-Refractory Sclerodermatous Chronic Graft-Versus-Host Disease (GVHD) With GDC-0449 (GDC-0449)
Brief Title: Vismodegib in Treating Patients With Steroid-Refractory Chronic Graft-Versus-Host Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02672; NCI-2014-02672 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IIT 9664; 84584; 9664 (Other: Huntsman Cancer Institute/University of Utah); 9664 (Other: CTEP); P30CA042014 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care (vismodegib) (Experimental): Patients receive vismodegib PO daily, every other day, every three days, or twice weekly for 6-12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Vismodegib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This pilot clinical trial studies how well vismodegib works in treating patients with chronic graft-versus-host disease that did not respond to previous steroid treatment. Chronic graft-versus-host disease can cause a build-up of scar tissue under the skin and lead to symptoms such as sclerodermatous skin changes, dry mouth, dry eye, narrowing of the esophagus, or vaginal graft-versus-host disease. Vismodegib may work against the build-up of scar tissue and be a better treatment for chronic graft-versus-host disease caused by a hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical effects of GDC-0449 (vismodegib), in steroid-refractory chronic graft-versus-host disease (GVHD).

SECONDARY OBJECTIVES:

I. To determine the safety of GDC-0449 in patients with steroid-refractory GVHD.

II. To determine the change in National Institutes of Health (NIH) Consensus Criteria (CC) global score of chronic GVHD at 6 and 12 months from baseline.

III. To determine one-year non relapse mortality (NRM) and one-year relapse rate.

IV. To determine one-year failure free survival (FFS) and one-year overall survival (OS).

V. To determine baseline clinical characteristics that may be associated with decreased FFS.

OUTLINE:

Patients receive vismodegib orally (PO) daily, every other day, every three days, or twice weekly for 6-12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 months
* Leukocytes >= 3,000/microliter (mcL)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 50,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT))/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 2.5 x institutional upper limit of normal
* Creatinine =< 1.5 mg/dl OR creatinine clearance >= 55 mL/min using the Cockcroft-Gault equation for patients with creatinine levels above 1.5 mg/dl
* Patients with chronic GVHD diagnosed within 3 years after hematopoietic stem cell transplant (HSCT) for any disease, with any graft, and any conditioning regimen with at least one manifestation secondary to fibrosis, including: sclerodermatous skin changes, dry mouth, dry eye, esophageal strictures, or vaginal GVHD
* Failure to respond to corticosteroids, defined as:

  * Progression of chronic GVHD despite optimal first line therapy (> 0.5 mg/kg/day of prednisone dose equivalent (PDE) for two weeks) or
  * No improvement after 4-8 weeks of sustained therapy; sustained therapy should include 2 weeks of > 0.5 mg/kg/day of PDE or
  * Inability to taper steroid dosage to less than 0.5 mg/kg/day of PDE without worsening of chronic GVHD or
  * Need for second or third line therapy beyond corticosteroids and calcineurin inhibitors or sirolimus, irrespective of other criteria
* Women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 24 months post-treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 milli-international unit (mIU)/mL) within 7 days prior to the first dose of GDC-0449 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of GDC-0449; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of GDC-0449 cause serious or life-threatening birth defects; patients must continue highly effective contraception during therapy and for 24 months after the last dose of GDC-0449
  * Women of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had a tubal ligation
  * Women are considered not to be of childbearing potential for the following reasons:

    * The patient has undergone hysterectomy and/or bilateral oophorectomy
    * The patient is post-menopausal defined by amenorrhea for at least 12 months in a woman > 45 years old
  * Male patients should use condoms with spermicide, even after a vasectomy, during sexual intercourse with female partners while being treated with GDC-0449 and for 3 months after the last dose to avoid exposing an embryo or fetus to GDC-0449
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are eligible provided that they meet the following criteria in addition to the other protocol criteria:

  * Cancer as the only acquired immunodeficiency syndrome (AIDS)-defining condition
  * Cluster of differentiation (CD)4 cell count >= 250
  * Treatment sensitive HIV and prospects for long term survival on the basis of HIV disease alone
  * Willing to take anti-HIV therapy that will have minimal potential for pharmacokinetic interactions with GDC-0449

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449
* Patients receiving any medications or substances that are strong inducers/inhibitors or substrates of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)/5, cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9), CYP2C8, or CYP2C19 are ineligible; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow capsules
* Patients with clinically important history of liver disease, including viral or other hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GDC-0449
* More than 2 lines of therapy beyond corticosteroids with or without calcineurin inhibitors or sirolimus
* Relapsed malignancy after transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Couriel, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Vismodegib)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.67 (12.16)
Age, Continuous [Median (Full Range); unit: years] | 53 [36 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Baseline Chronic GVHD Grade [Count of Participants; unit: Participants] — Chronic graft-versus-host disease (GVHD) severity was assessed with the National Institutes of Health (NIH) global score of chronic GVHD, which was defined using the 2014 NIH consensus criteria for diagnosis and staging of chronic GVHD. This system stages severity in each individual organ, and then reports a global score defined as mild, moderate or severe, based on number of organs involved and organ severity score.
  Participants
    Mild GVHD | 0
    Moderate GVHD | 0
    Severe GVHD | 6

OUTCOME MEASURES:

1. Primary Outcome: Failure Free Survival (FFS)
Description: Defined as the count of participants at six months with an absence of non relapse mortality (NRM), no recurrent malignancy, steroid dose at 6 months =< 0.2 mg/kg/day of prednisone dose equivalent (PDE), and no addition of new systemic treatment for chronic graft-versus-host disease (GVHD) at six months after start of treatment.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Participants | 3

2. Secondary Outcome: Incidence of Adverse Events
Description: The count of participants who experience adverse events (AE) and serious adverse events (SAE) while on treatment or within one month after discontinuing treatment.
Time Frame: Up to 1 month post last date of treatment (max time of approximately one year)
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Participants
  Participants with any AE | 6
  Participants with any SAE | 4

3. Secondary Outcome: Chronic Graft-versus-host Disease Response
Description: Chronic graft-versus-host disease (GVHD) severity was assessed at baseline with the National Institutes of Health (NIH) global score of chronic GVHD, which was defined using the 2014 NIH consensus criteria for diagnosis and staging of chronic GVHD (see Baseline Characteristics). Following initiation of treatment, the response to therapy was assessed as complete response (CR) (complete resolution of GVHD in one or more organ system) , partial response (PR) (improvement of GVHD in one or more organ system), stable disease (SD) (no change in GVHD), or progressive disease (PD) (worsened GVHD in one or more organ system), based on 2014 NIH consensus criteria for response assessment. GVHD was assessed monthly, with defined study endpoints at 6 and 12 months. Additionally, best overall response on the study is being reported to include response for patients who did not remain on study long enough to be included in the 6 month assessment.
Time Frame: Baseline to up to 12 months after initiation of protocol therapy
Population: Only 3 participants had NIH GVHD assessment for response at 6 months. Only 1 participant had NIH GVHD assessment for response at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Participants
  Best Overall Response on study: Partial Response (PR) | 6
  Best Overall Response on study: CR, SD, and PD | 0
  Response at 6 months: number analyzed (Participants) | 3
  Response at 6 months: Partial Response (PR) | 3
  Response at 6 months: CR, SD, and PD | 0
  Response at 12 months: number analyzed (Participants) | 1
  Response at 12 months: Partial Response (PR) | 1
  Response at 12 months: CR, SD, and PD | 0

4. Secondary Outcome: One-year Non Relapse Mortality (NRM)
Description: Relapse will be defined as malignancy relapse or as the initiation of any unintended intervention including an unplanned taper of immunosuppressant therapy to prevent malignancy progression due to any signs of recurrent, residual or new malignant disease after transplantation. Non relapse mortality is the number of participant deaths due to any cause other than relapse.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Participants | 0

5. Secondary Outcome: One Year Relapse
Description: Relapse will be defined as malignancy relapse or as the initiation of any unintended intervention including an unplanned taper of immunosuppressant therapy to prevent malignancy progression due to any signs of recurrent, residual or new malignant disease after transplantation. This measure is reported as the count of participants who experienced a relapse of their primary malignancy within one year of starting study therapy.
Time Frame: Up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Participants | 1

6. Secondary Outcome: One-year Failure Free Survival (FFS)
Description: Defined as the count of participants at one year with an absence of non relapse mortality (NRM), no recurrent malignancy, steroid dose at 6 months =< 0.2 mg/kg/day of prednisone dose equivalent (PDE), and no addition of new systemic treatment for chronic graft-versus-host disease (GVHD) at one year after start of treatment.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Participants | 1

7. Secondary Outcome: One-year Overall Survival
Description: A count of participants who are not deceased at one year after initiation of study therapy.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Participants | 5

8. Secondary Outcome: Clinical Characteristics Associated With Failure Free Survival (FFS)
Description: The study proposed to evaluate clinical characteristics that could be associated with FFS. Each patient was categorized as either having FFS greater than 6 months or less than 6 months. Factors evaluated were whether or not the patient had high intensity conditional with total-body irradiation (TBI) before bone marrow transplant, whether or not the patient had > 3 involved sites with chronic graft versus host disease (GVHD), whether or not the patient had lower gastrointestinal (GI) involvement by GVHD, and whether or not the patient had a Severe NIH global score at initiation of protocol treatment.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Vismodegib)
Number analyzed (Participants) | 6
Participants
  Factor: TBI before transplanat: Had Factor and FFS > 6 months | 1
  Factor: TBI before transplanat: Did not have factor and FFS > 6 months | 2
  Factor: TBI before transplanat: Had factor and FFS < 6 months | 1
  Factor: TBI before transplanat: Did not have factor and FFS < 6 months | 2
  Factor: Greater than 3 sites involved with GVHD: Had Factor and FFS > 6 months | 1
  Factor: Greater than 3 sites involved with GVHD: Did not have factor and FFS > 6 months | 2
  Factor: Greater than 3 sites involved with GVHD: Had factor and FFS < 6 months | 2
  Factor: Greater than 3 sites involved with GVHD: Did not have factor and FFS < 6 months | 1
  Factor: Lower GI involvement with GVHD: Had Factor and FFS > 6 months | 2
  Factor: Lower GI involvement with GVHD: Did not have factor and FFS > 6 months | 1
  Factor: Lower GI involvement with GVHD: Had factor and FFS < 6 months | 2
  Factor: Lower GI involvement with GVHD: Did not have factor and FFS < 6 months | 1
  Factor: Severe NIH Global GVHD Score: Had Factor and FFS > 6 months | 3
  Factor: Severe NIH Global GVHD Score: Did not have factor and FFS > 6 months | 0
  Factor: Severe NIH Global GVHD Score: Had factor and FFS < 6 months | 3
  Factor: Severe NIH Global GVHD Score: Did not have factor and FFS < 6 months | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment until 30 days after the last dose, up to one year.
Description: The occurrence of adverse events (AEs) was sought by non-directive questioning of the patient at each visit or phone contact during the study. Adverse events may also have been detected when they were volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments.
Arm/Group | Supportive Care (Vismodegib)
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Vismodegib) (N=6)
Fracture (Injury, poisoning and procedural complications) | 1
Hypotension (Vascular disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumatosis (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1 (2)
Weight loss (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Vismodegib) (N=6)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Agitation (Psychiatric disorders) | 1
Alkaline phosphatase increased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 (7)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
BUN elevated (Metabolism and nutrition disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
colonic polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Concentration impairment (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
conjunctival irritation lower eye (Eye disorders) | 1
Coronary atherosclerosis (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 1
crown of tooth detached (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 4 (7)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
elevated neutrophils (Blood and lymphatic system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Epstein Barr Virus (Infections and infestations) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Flu like symptoms (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 2
Gastritis (Gastrointestinal disorders) | 1
gastrointestinal disorder (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Increased Appetite (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 2 (3)
leg ulceration (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
Movements involuntary (Nervous system disorders) | 3 (6)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 5
Neutrophil count decreased (Investigations) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis infective (Infections and infestations) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Spasticity (Nervous system disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2 (3)
Vasculitis (Vascular disorders) | 1
Weight loss (Investigations) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT02337517/Prot_SAP_000.pdf